CLINICAL TRIAL: NCT07150650
Title: Exploring Novel Biomarkers of ICU-AW in Mechanically Ventilated Children at the Molecular Level
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ICU-AW 20250821
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: ICU Acquired Weakness
Keywords: ICU Acquired Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Collection: From the residual blood of routine tests, 3 mL of EDTA-anticoagulated whole blood was collected and centrifuged at 3000 × g for 15 minutes (4°C).
  Aliquoting and Storage: The supernatant was aliquoted into 500 μL cryovials and stored in a -80°C ultra-low temperature freezer (temperature fluctuation < ±2°C).
  Time Points: Day 0 (upon enrollment), Day 3 (acute phase), Day 7 (progressive phase), and Day 10 (recovery phase/outcome assessment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU-AW: Children receiving mechanical ventilation who developed ICU-AW at the study endpoint.
  Interventions: Diagnostic Test: ICU-AW
- without ICU-AW: Children receiving mechanical ventilation who did not developed ICU-AW at the study endpoint.

INTERVENTIONS:
Diagnostic Test: ICU-AW — The enrolled children receiving mechanical ventilation were grouped based on the occurrence of ICU-acquired weakness (ICU-AW) at the study endpoint.
  Groups: ICU-AW

SUMMARY:
Acquired weakness (AW) is a common complication among patients in the Intensive Care Unit (ICU). It is a systemic muscle weakness and dysfunction associated with critical illness, often related to prolonged bed rest, mechanical ventilation, systemic inflammatory response syndrome (SIRS), and multiple organ dysfunction syndrome (MODS). The primary clinical manifestations include weakness in limb and respiratory muscles, particularly diminished strength in distal muscle groups. As a result, the weaning process from mechanical ventilation becomes more challenging, leading to prolonged ICU stays, increased mortality, and a higher risk of long-term functional disability. The significance of AW lies not only in its substantial impediment to short-term recovery but also in its role as a core component of Post-Intensive Care Syndrome (PICS), profoundly affecting patients' long-term outcomes.

Mechanical ventilation is a vital life-support technology for critically ill children in the Pediatric Intensive Care Unit (PICU). However, complications associated with mechanical ventilation have garnered increasing attention, particularly Acquired Weakness in mechanically ventilated children. With improving survival rates in the PICU, a growing number of pediatric critical illness survivors are at risk of developing AW. Despite rapid advancements in pediatric critical care medicine in China, there is currently a lack of an early warning system for AW in children receiving mechanical ventilation, resulting in significantly delayed clinical interventions. This project aims to identify novel biomarkers for pediatric ICU-AW and develop an early warning model. It holds promise for transitioning from the traditional post-symptomatic diagnostic approach to subclinical prediction of AW in children, which is of great clinical value for reducing disability rates and optimizing critical care rehabilitation strategies.

DETAILED DESCRIPTION:
An electronic database was established to collect clinical data from mechanically ventilated children, including baseline clinical characteristics, laboratory test results, and imaging data. Each participating research center designated dedicated investigators to enroll study subjects starting on the same date (eligible patients already hospitalized on the start date were included). These investigators were responsible for data cleaning, organization, and standardization to ensure data quality. For all enrolled patients, data on demographic characteristics, clinical features, and laboratory test results were recorded using case report forms (CRFs) on the day of enrollment (D0), day 3 (D3), day 10 (D10), the day of discharge from the pediatric intensive care unit (Ddis), or the day of death (DD).

To investigate the pathophysiology of ICU-acquired weakness (ICU-AW) under the inflammation-metabolism-neuromuscular injury hypothesis, dynamic plasma biological sample collection was performed. Samples were collected at different time points during mechanical ventilation to establish a biobank. Proteomic and genomic multi-omics approaches were employed to screen for inflammatory cytokines, specific degradation biomarkers of muscle injury, and metabolism-related genes such as those involved in mitochondrial function. Levels of these biomarkers in biological samples from mechanically ventilated children were measured to analyze their association with the onset and progression of ICU-AW, thereby untangling the pathophysiology of ICU-AW at the molecular level.

The Pathophysiology of ICU-AW remains unclear, and there is a lack of research exploring its molecular mechanisms, making it difficult to identify effective early warning indicators. Currently, it is believed that the pathophysiology of ICU-AW is associated with persistent inflammation, immunosuppression, and catabolic syndrome (PICS), resulting from the interplay of multiple factors and pathways. Key mechanisms include: inflammatory response and immune dysregulation, mitochondrial dysfunction and abnormal energy metabolism, oxidative stress, and microvascular changes, which collectively lead to muscular and neurological dysfunction. The core of its pathophysiology lies in the imbalance between protein synthesis and muscle protein degradation, which occurs in response to various stimuli. Key mechanisms include: 1) The ubiquitin-proteasome system (UPS). Pro-inflammatory cytokines (e.g: NF-κB) upregulate muscle-specific E3 ubiquitin ligases (such as MuRF1 and Atrogin-1), accelerating muscle protein degradation and contributing to muscle atrophy. 2) The autophagy-lysosome system. Abnormal activation of this system leads to muscle fiber atrophy, though its specific regulatory mechanisms remain unclear. Although some progress has been made in mechanistic studies of ICU-AW, its pathophysiological mechanisms are complex and not yet fully elucidated. There is a lack of biomarkers for early clinical identification and insufficient translational molecular research.

In recent years, the discovery of multi-dimensional molecular markers has provided new directions for early identification and mechanistic analysis of ICU-AW:

1. Direct markers of muscle structural damage: Urinary Titin. As a core protein of the muscle cytoskeleton, its release in urine quantitatively reflects the extent of muscle fiber breakdown. The mechanism of its release is closely related to key pathological pathways of ICU-AW (UPS activation, inflammation-oxidative stress synergy, and dysregulated mechanical signaling). A multicenter prospective study found that urinary Titin levels in non-surgical ICU patients were 10 to 30 times higher than normal levels and were significantly negatively correlated with dynamic changes in rectus femoris cross-sectional area measured by ultrasound (p < 0.01), suggesting its potential as a non-invasive biomarker for monitoring muscle atrophy.
2. Combined markers of neuromuscular interaction damage: Neurofilament light chain (NfL)-a major cytoskeletal protein of neuronal axons and a marker of axonal injury-was significantly elevated in the serum of ICU-AW patients with CIP/CIM early after admission (median 4 days); Glial fibrillary acidic protein (GFAP)-reflecting astrocyte activation-contributes to the onset and progression of ICU-AW by mediating neuroinflammation, motor neuron injury, and neuromuscular junction dysfunction. Their dynamic changes not only offer new tools for early diagnosis and prognosis assessment of ICU-AW but may also represent potential targets for future therapeutic interventions.
3. Epigenetic regulatory markers: Abnormal DNA methylation and muscle dysfunction. HIC1 regulates muscle regeneration and modulates the concentration of postsynaptic acetylcholine receptors, while NADK2 is involved in lipid metabolism and mitochondrial stimulation. Recent studies in adults have shown that, compared to controls, ICU patients exhibit reduced methylation in the epigenomic regions of HIC1 and NADK2. The HIC1 and NADK2 genes may theoretically provide a biological basis for ICU-AW.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 28 days and 18 years;
2. Patients continuously admitted to the PICU during the study period and subjected to invasive mechanical ventilation.

Exclusion Criteria:

1. Mechanical ventilation duration < 72 hours;
2. Presence of primary central or neuromuscular diseases that significantly affect central or peripheral respiratory failure, including: traumatic brain injury, cerebrovascular disease history (e.g., cerebral hemorrhage, cerebral infarction), intracranial tumors, central nervous system infections, spinal cord injury, Guillain-Barré syndrome, porphyria, paraneoplastic neuropathy, etc.;
3. Conditions requiring immobilization such as limb joint surgery or fractures.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Age between 28 days and 18 years;
  2. Patients continuously admitted to the PICU during the study period and subjected to invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence rate of ICU-AW | Diagnosis of ICU-AW in mechanically ventilated children was determined based on assessments at day 10.
  The occurrence rate of ICU-AW in mechanically ventilated children on day 10. ICU-AW was defined as: MRC score < 48, or slowed nerve conduction velocity on electromyography; CIP: normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, reduced mixed SNAP amplitude; CIM: normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, decreased muscle excitability to direct stimulation, increased CMAP duration, normal SNAP; or confirmed by muscle biopsy.
expression changes of differential proteins | Proteomic analyses were performed on blood samples collected on day 3 and day 10.
  Data Processing: Data preprocessing, peak identification in mass spectra, noise reduction, and quantitative analysis were performed using Bruker's Spectronaut or other relevant software. The use of Data-Independent Acquisition (DIA) technology enabled the acquisition of unbiased quantitative data.
  Differential Protein Screening: Differential analysis was conducted on the obtained protein data to identify proteins that exhibited significant changes between the acquired weakness group and the control group. Statistical methods (such as t-test and ANOVA) were applied to analyze the data and determine expression changes of differential proteins.
  Functional Enrichment Analysis: Pathway enrichment analysis was carried out using databases (e.g., GO, KEGG, Reactome) to explore biological pathways and molecular mechanisms associated with acquired weakness.
Differential Metabolite Analysis | Metabolomic analyses were performed on blood samples collected on day 3 and day 10.
  Differential Metabolite Analysis: Statistical methods (e.g., t-test, ANOVA, etc.) were employed to analyze differences in metabolite abundance among different experimental groups, aiming to identify metabolites that exhibited significant changes under varying conditions.
  Metabolic Pathway Analysis: Pathway enrichment analysis was performed using bioinformatics tools (e.g., MetaboAnalyst, Ingenuity Pathway Analysis, etc.) to untangle potential biological mechanisms associated with the altered metabolites.
  Multivariate Analysis: Multivariate analytical approaches, including principal component analysis (PCA) and partial least squares-discriminant analysis (PLS-DA), were applied to conduct cluster analysis of the experimental data and to discern metabolite pattern differences between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Children' hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banwell BL, Mildner RJ, Hassall AC, Becker LE, Vajsar J, Shemie SD. Muscle weakness in critically ill children. Neurology. 2003 Dec 23;61(12):1779-82. doi: 10.1212/01.wnl.0000098886.90030.67. PMID 14694046
- [Background] Zhang Z, Tao J, Cai X, Huang L, Liu C, Ren H, Qu D, Gao H, Cheng Y, Zhang F, Yang Z, Xu W, Miao H, Liu P, Liu Y, Lu G, Chen W. Clinical characteristics and outcomes of children with prolonged mechanical ventilation in PICUs in mainland China: A national survey. Pediatr Pulmonol. 2023 May;58(5):1401-1410. doi: 10.1002/ppul.26332. Epub 2023 Feb 8. PMID 36705329
- [Background] Zhang Z, Cai X, Ming M, Huang L, Liu C, Ren H, Qu D, Gao H, Cheng Y, Zhang F, Yang Z, Xu W, Miao H, Liu P, Liu Y, Lu G, Chen W. Incidence, outcome, and prognostic factors of prolonged mechanical ventilation among children in Chinese mainland: a multi-center survey. Front Pediatr. 2024 May 30;12:1413094. doi: 10.3389/fped.2024.1413094. eCollection 2024. PMID 38873585
- [Background] Johnson RW, Ng KWP, Dietz AR, Hartman ME, Baty JD, Hasan N, Zaidman CM, Shoykhet M. Muscle atrophy in mechanically-ventilated critically ill children. PLoS One. 2018 Dec 19;13(12):e0207720. doi: 10.1371/journal.pone.0207720. eCollection 2018. PMID 30566470
- [Background] Kalb R. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Jul 17;371(3):287. doi: 10.1056/NEJMc1406274. No abstract available. PMID 25014704